CLINICAL TRIAL: NCT03361839
Title: Clinical Trail for Study Endometrial Receptivity in RIF
Brief Title: Endometrial Receptivity in Patients With Recurrent Implantation Failure as a Preparatory Step for PET
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Nooh Riad Ali, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: example -1
Record Dates: First submitted 2017-11-18; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: RIF , Endometrial Receptivity

STUDY DESIGN:
Intervention Model Description: non randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): patients with RIF
  Interventions: Diagnostic Test: endometrial biopsy
- 2 (Placebo Comparator): fertile arm as r reference for result
  Interventions: Diagnostic Test: endometrial biopsy

INTERVENTIONS:
Diagnostic Test: endometrial biopsy — endometrial biopsy for genetic study of endometrial receptivity

SUMMARY:
clinical trial to improve pregnancy outcome in patient with RLF , study done on 2 phases. phase 1 to study variations of endometrial receptivity genes in this group of patient, phase 2 repeat cycle or transfer frozen embryo in proper time and after giving proper treatment

DETAILED DESCRIPTION:
Study design: Nonrandomized clinical trial

Inclusion criteria: women with history of recurrent implantation failure with History of transfer of at least 4 good quality embryos in at least 3 fresh or frozen cycles

* Women age less than 40 years

  * BMI (25 - 33)
  * Non diabetic Arms of study: 2

    1. Women for frozen embryo transfer or New ICSI cycle fulfilling previous criteria (study arm).
    2. Control group of fertile patient (fertile patients receiving local mechanical contraception as a reference group). To help in identification of cut off values of all related genes.

       Sample size: 60 Intervention

       Phase 1

    <!-- -->

    1. Recent labs ( day 2 serum FSH,LH TSH , PROLACTIN serum E 2)within 6 ms
    2. White tablets of cycloprogenova 4 mg /12 hs twice / day
    3. Add progesterone on (day 9) 600 mg per day.
    4. On day 5 of start progesterone do endometrial biopsy using pipplle endometrial suction curette
    5. Indirect immunofluorescence using QRT-PCR of the endometrial tissue for 11 genes necessary for implantation and maintenance of pregnancy. Classify EB as pre-receptive, receptive and post receptive and plan next day of transfer.
    6. Genes to be studied: the most accessible genes will be studied.

    <!-- -->

    1. Homeobox gene (HOXA-10 ) upregulated
    2. LIF upregulated
    3. Alpha VB3 integren and its ligand osteopontin are positively detected
    4. ECM upregulated
    5. Paracrine stromal factors, +ve (EGF (epidermal growth factor), heparin binding EGF)
* VE 17 B estradiol (E2 factors) 6- L selectin upregulated 7- E-cadherin ( downregulated) 8- Intercellular cell adhesion molecules highly expressed 9- Mucin 1 down regulated at implantation 10- IL-6 upregulated 11- IL-1 and IL- 1 R upregulated 12- Prostaglandin transporter (PGT) reduced in mid-late secretory. Phase 2 7- In the study arm Next cycle start active ttt cycle of frozen ET( white tablet of Cycloprogenova twice daily then at day 9 do transvaginal US when endometrial thickness is more than 9 mm start progesterone till day 5 for transfer of frozen embryos or new ICSI cycle according to standard protocol ( long or antagonist protocols according to every patient data ). then select one of the suggested treatment

  1. Intrauterine injection of human chorionic gonadotropins before transfer
  2. Granulocyte colony stimulating factor given intrauterine ( 300 mcg /ml on day of OP or progesterone administration of FET
  3. Recombinant LIF
  4. Or combination of 1 and 2 Common measures to be done in any situation

  <!-- -->

  1. Low dose aspirin 75 mg daily
  2. Steroids 5 mg hostacortin daily
  3. Endometrial injury cycle before active cycle treatment

  8- Technique of QRT-PCR of endometrial receptivity genes RNA Extraction Cells of all studied groups will be lysed and total RNA was isolated with RNAeasy Mini Kit (Qiagen) and further analyzed for quantity and quality with Beckman dual spectrophotometer (USA).

Real Time PCR (qRT-PCR) For quantitative expression of HOXA-10, LIF, Alpha VB3 integren and its ligand osteopontin, ECM, EGF, E2 FACTOR, L-selectin, E-cadherin, ICAM, Mucin1, IL-6, IL1, IL-1R and PGT; the following procedure will bes assessed. 10 ng of the total RNA from each sample will be used for cDNA synthesis by reverse transcription using High capacity cDNA Reverse Transcriptase kit (Applied Biosystem, USA). The cDNA will be subsequently amplified with the Syber Green I PCR Master Kit (Fermentas) in a 48-well plate using the Step One instrument (Applied Biosystem, USA) as follows: 10 minutes at 95 ºC for enzyme activation followed by 40 cycles of 15 seconds at 95ºC, 20 seconds at 55 ºC and 30 second at 72 ºC for the amplification step. Changes in the expression of each target gene will be normalized relative to the mean critical threshold (CT) values of β-actin as housekeeping gene by the ΔΔCt method. We will use 1 μM of both primers specific for each target gene. DNA sequencing will be assessed for all studied genes

ELIGIBILITY:
Inclusion Criteria:

* women with history of recurrent implantation failure with History of transfer of at least 4 good quality embryos in at least 3 fresh or frozen cycles
* Women age less than 40 years • BMI (25 - 33)

Exclusion Criteria:

* diabetic women

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | two weeks after transfer
  positive intrauterine sac

CONTACTS AND LOCATIONS:
Overall Officials: abdelmegeed ramzy, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No
net results data

REFERENCES:
- [Background] Nejat EJ, Ruiz-Alonso M, Simon C, Meier UT. Timing the window of implantation by nucleolar channel system prevalence matches the accuracy of the endometrial receptivity array. Fertil Steril. 2014 Nov;102(5):1477-81. doi: 10.1016/j.fertnstert.2014.07.1254. Epub 2014 Sep 17. PMID 25241377